CLINICAL TRIAL: NCT02624479
Title: Phase I Pharmacokinetic Pilot Study to Investigate the Bioavailability and Tolerability of Three Different Oral Formulations of Sodium Thiosulfate
Brief Title: Pharmacokinetic Study to Investigate the Bioavailability and Tolerability of 3 Oral Formulations of Sodium Thiosulfate
Acronym: TSTS
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Formulations could never be successfully produced
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 009_15
Record Dates: First submitted 2015-11-26; First posted 2015-12-08 (Estimated); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Healthy
Keywords: Pharmacokinetics
MeSH Terms: interventions — sodium thiosulfate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fast first (Experimental): Sodium thiosulfate fast release formulation first, followed by medium and slow
  Interventions: Drug: Sodium thiosulfate
- Medium first (Experimental): Sodium thiosulfate medium release formulation first, followed by slow and fast
  Interventions: Drug: Sodium thiosulfate
- Slow first (Experimental): Sodium thiosulfate slow release formulation first, followed by fast and medium
  Interventions: Drug: Sodium thiosulfate

INTERVENTIONS:
Drug: Sodium thiosulfate — oral administration of thiosulfate

SUMMARY:
Chronic treatment and prophylaxis of vessel and soft tissue calcification as well as of renal calculi could be a future indication for sodium thiosulfate (STS). Using an oral formulation might increase the compliance and treatment success compared to parenteral administration.

Three gastro-resistant formulations of STS for oral administration were developed with different release characteristics: fast-release, medium-release and slow-release tablets. Aim of the enteric coating was to increase the oral bioavailability of STS. The bioavailability and tolerability of these formulations for oral administration in healthy volunteers will be compared in this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female healthy subjects ≥ 18 years
* Negative pregnancy test in female subjects of childbearing age
* Able to understand character and individual consequences of the clinical trial and to provide written informed consent to participate in the study

Exclusion Criteria:

* Pregnant or lactating subjects.
* Renal impairment (creatinine clearance <60ml/min)
* Concomitant medication
* Gastrointestinal diseases
* History of alcohol abuse, illicit drug use, significant mental illness, physical dependance to opioid, other drug abuse or addiction (last 12 months)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Relative bioavailability of STS after oral administration based on urinary excretion of TS and sulfate | 7 weeks

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | 7 weeks
TS excretion in urine | 48 hours
  amount excreted within 48h and fraction (amount/dose) of administered thiosulfate
TS excretion in urine: amount | 48 hours
  amount excreted within 48h
TS excretion in urine: fraction of administered TS | 48 hours
  excreted / administered
Sulfate excretion in urine: amount | 48 hours
  amount excreted within 48h
Sulfate excretion in urine: fraction of administered TS | 48 hours
  excreted / administered

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Uehlinger, Prof Dr.med., Study Chair — Insel Gruppe AG, University Hospital Bern